CLINICAL TRIAL: NCT02543190
Title: System-Wide Improvement for Transitions After Surgery: The SWIFT Post op Program
Acronym: SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Colon and Rectal Surgery Associates, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1408M52923
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Colectomy; Colorectal Surgery; Ileostomy
Keywords: Care Transition; Readmission; Rehospitalization

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider did not know study assignment. Reviewer for primary outcomes did not know study assignment
Oversight: Data Monitoring Committee: No

ARMS (2):
- compliance surveillance (Experimental): * Prospective audits by study personnel
  * Call from the clinic nurse practitioner or physician's assistant within 7 days of discharge to administer a screening questionnaire to identify patients at risk of dehydration. Study personnel will ensure this phone call is made.
  Interventions: Behavioral: compliance surveillance and improvement strategy
- Usual Care (No Intervention): educational session at the start of the study

INTERVENTIONS:
Behavioral: compliance surveillance and improvement strategy — External monitor to ensure compliance with an educational protocol.
  Arms: compliance surveillance

SUMMARY:
Short-term post-operative complications after colon and rectal surgery present a known major clinical and financial burden for patients and hospitals. Focused efforts to reduce readmissions after colorectal surgery is one potentially high-yield and broad approach to address this problem since post- operative complications are the strongest predictor of readmissions. We focus on decreasing readmissions after ileostomy surgery by using a previously published intervention that prevents dehydration in the outpatient setting and decreases acute renal failure complications. We plan to introduce the SWIFT post op program for ileostomy patients at one academic and two community hospitals which are part of a single health care system, and to then randomize patients to usual care in the setting of this new program versus an aggressive compliance surveillance and improvement strategy (CSIS) strategy using study personnel. Our primary study outcome is all-cause 30-day readmission, and our secondary outcomes include patient satisfaction (CAHPS scores) and a cost-benefit analysis. We seek to create a partnership between colorectal surgeons, inpatient nurse managers and wound ostomy continence nurses (WOCN) at the three sites, linking them with outpatient nurse practitioners and physician's assistants at the respective colorectal surgery clinics who facilitate care-transition after hospital discharge.

DETAILED DESCRIPTION:
At the start of the study, inpatient and outpatient nurses, physicians and physicians assistants will be oriented to the intervention in the study and will be suggested that the intervention is standard of care based on the following study:

Nagle D, Pare T, Keenen E, Marcet K, Tizio S, Poylin V*. Ileostomy Pathway Virtually Eliminates Readmissions for Dehydration in New Ostomates. Diseases of the Colon and Rectum 2012; 55: 1266-1272.

The intervention patients will be subject to a compliance surveillance and intervention strategy (CSIS) administered by study personnel to encourage the following and persist with telephone calls if the following have not been achieved.

* Prospective audits by study personnel to check and encourage teaching in the clinic, teaching on the wards, and telephone follow up occurred.
* A self-assessment tool for patients and families to confirm understanding of the education materials.
* Coaching of inpatient nurses taking care of ileostomy patients by WOCN and/or the inpatient nurse champion
* Call from the clinic nurse practitioner or physician's assistant within 7 days of discharge to review the educational materials and administer a screening questionnaire to identify patients at risk of dehydration. In patients randomized to CSIS, study personnel will ensure this phone call is made.

The usual care arm will include no such surveillance.

The randomized study will be powered to detect a decrease in hospital readmission rates (all-cause) from 25% to 5%. Secondary outcomes include readmission due to dehydration and patient satisfaction (Surgical-CAHPS survey)

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled or who undergo ileostomy alone or as part of a multiple procedure operation
* patients who have had an ileostomy in the past are eligible
* patients who have an ileostomy to address a recent surgical complication are eligible

Exclusion Criteria:

* Patients who have an ileostomy already in place immediately prior to the procedure (ie. revision, transposition, or parastomal hernia procedures
* patients on dialysis
* patients who require chronic TPN, IVF, or have short gut
* non-English speaking patients who do not have easy access to an appropriate interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Readmission to the hospital | 30 days after hospital discharge

SECONDARY OUTCOMES:
Patient satisfaction | 3-6 months after surgery
  S-CAHPS
Index length-of-stay | Index length-of-stay
  Time from surgical date to hospital discharge
Emergency room visit | 30 days after hospital discharge
  Emergency room visits for any reason 30 days after surgery
Total hospital-length-of-stay | 30 days after hospital discharge
  Total hospital length of stay for any reason after surgery
Readmission due to dehydration or acute renal failure | 30 days after hospital discharge
  Dehydration by clinician assessment, acute renal failure defined as elevation in creatinine to >2 mg/dl, or oliguria/anuria
Post-discharge follow up phone call | 30 days after hospital discharge
  Nurse, physician, or physician-assistant documentation of phone call to the patient that describes monitoring of ileostomy output volume

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Kwaan, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Medical Center -Fairview, Minneapolis, Minnesota
  - Colon and Rectal Surgery Associates, Saint Paul, Minnesota